CLINICAL TRIAL: NCT07337876
Title: Organ Preservation in Rectal Cancer by Dose Escalated MR Guided Adaptive Radiotherapy
Acronym: MARS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Cihan Gani, Prof., University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 311/2025BO1
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
Keywords: organ preservation
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR guided dose escalated radiotherapy (Experimental): A dose of 65 Gy is delivered to the primary tumor and affected lymph nodes.
  Interventions: Radiation: Dose escalated radiotherapy using a 1.5 T MR-Linac

INTERVENTIONS:
Radiation: Dose escalated radiotherapy using a 1.5 T MR-Linac — Dose escalated radiotherapy using a 1.5 T MR-Linac is given to the primary tumor and affected lymph nodes in an online adaptive manner

SUMMARY:
This study is testing whether radiation delivered with MRI guidance using a so-called MR-linac in distal rectal cancer can result in a high rate of organ preservation. Patients will receive radiotherapy together with standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of rectal cancer localized between dentate line and 12 cm from the anocutaneous line
* Any MRI staged rectal cancer meeting the following criteria
* cT1-cT3 and
* cN0 -cN1 and
* cM0
* Inclusion of UICC Stage I tumors only if unsuitable for endoscopic resection or if primary surgery would require permanent colostomy or deep anastomosis with expected poor organ function.
* Tumor affects less than 70% of the rectal circumference.
* Maximum longitudinal extension of the tumor less than 8 cm on MRI
* MR-Staging requirements: High-resolution, thin-sliced (i.e.

  ≤3mm) magnetic resonance imaging (MRI) of the pelvis.
* Cross-sectional imaging of the abdomen and chest to exclude distant metastases.
* Aged at least 18 years. No upper age limit.
* WHO/ECOG Performance Status ≤ 1
* Adequate hematological, hepatic, renal and metabolic function parameters
* Informed consent of the patient

Exclusion Criteria:

* Lower border of the tumor localised more than 12 cm from the anocutaneous line as measured by rigid rectoscopy
* Distant metastases
* Preexisting fecal incontinence for solid stool
* Prior antineoplastic therapy for rectal cancer
* Prior radiotherapy of the pelvic region
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidal jelly).
* Other concomitant antineoplastic therapy
* Serious concurrent diseases, including neurologic or psychiatric disorders (incl. dementia and uncontrolled seizures), active,uncontrolled infections, active, disseminated coagulation disorder
* Other primary tumors with an estimated life expectancy of less than three years
* Contraindications for treatment with 5-Fluorouracil or Capecitabine
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule (these conditions should be discussed with the patient before registration in the trial).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Two year TME-free survival | Two years from the start of radiotherapy
  Patients alive and without TME-surgery

SECONDARY OUTCOMES:
Clincal complete response rate | three months after the end of radiotherapy
  Patients who have no evidence of residual tumor on MRI and rectoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared if a sound scientific proposal if provided.